CLINICAL TRIAL: NCT00437723
Title: An Open-Label Study to Investigate the Effect of NeoRecormon on Hemoglobin Level and Renal Function in Patients With Chronic Kidney Disease, Stage 2-4
Brief Title: A Study of NeoRecormon in Patients With Chronic Kidney Disease.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20200
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: epoetin beta [NeoRecormon]
- 2 (No Intervention)

INTERVENTIONS:
Drug: epoetin beta [NeoRecormon] — At a dose to achieve and maintain an Hb level of 120-135g/dL.
  Arms: 1

SUMMARY:
This 2 arm study will compare the level of anemia, and the decline in renal function, between patients receiving NeoRecormon, and those not receiving it. Patients with chronic kidney disease, stage 2-4, and not receiving dialysis, will be randomized 2:1 to a group receiving NeoRecormon (at a dose determined by the investigator to achieve and maintain an Hb level of 120-135 g/L), or to a control group not receiving NeoRecormon. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients,18-75 years of age;
* end-stage renal disease, not on dialysis;
* Hb <110g/L.

Exclusion Criteria:

* unstable hypertension;
* acute infections;
* use of i.v. NeoRecormon, or use of any other ESA beside NeoRecormon;
* myocardial infarction, unstable angina or venous thrombosis within 6 months before start of treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Hb level, decline in renal function, 24h proteinuria, creatinine clearance. | Throughout study

SECONDARY OUTCOMES:
SAEs, AEs leading to withdrawal, AEs related to NeoRecormon. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Serbia (2):
  - Belgrade
  - Novi Sad